CLINICAL TRIAL: NCT04305782
Title: NIH Release/Relock Socket
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Joan Sanders, Professor, Department of Bioengineering, University of Washington
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006874; 2R01HD060585-08 (NIH)
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Lower Limb Amputation Below Knee (Injury)
Keywords: Prosthetic Socket; Amputee; Pin Lock Prosthetic Socket
MeSH Terms: conditions — Wounds and Injuries | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Release/Relock Socket - In Lab (Experimental): The test socket will be operated by the participant in lab, following a structured protocol. This arm focuses on the order effects on the re-lock panel and pin mechanisms on limb volume.
  Interventions: Device: Release/Relock Socket - In Lab
- Release/Relock Socket - Out of Lab (Experimental): The test socket will be operated by the participant out of lab, with no structured protocol. This arm focuses on the effects of the re-lock panel and pin mechanisms on participant comfort.
  Interventions: Device: Release/Relock Socket - Out of Lab
- Release/Relock Socket & Control (Experimental): The test socket will be operated by the participant out of lab, with no structured protocol. This arm focuses on the comparing participant experience using the novel mechanism versus traditional socket mechanisms.
  Interventions: Device: Release/Relock Socket - In Lab; Device: Release/Relock Socket & Control

INTERVENTIONS:
Device: Release/Relock Socket - In Lab — The participants will operate the test socket in one of two test conditions: (1) pin re-lock before panel re-lock and (2) panel re-lock before pin re-lock. Participants will test each of the two conditions in a random order, in lab, following a structured protocol. Tests will determine if the order of the re-lock mechanisms influences changes in limb volume.
  Arms: Release/Relock Socket & Control; Release/Relock Socket - In Lab
Device: Release/Relock Socket - Out of Lab — The participants will operate the test socket in one of two test conditions: (1) pin re-lock before panel re-lock and (2) panel re-lock before pin re-lock. Participants will test each of the two conditions in a random order, out of lab, with no structured protocol. Tests will determine if the order of the re-lock mechanisms changes participant experience.
  Arms: Release/Relock Socket - Out of Lab
Device: Release/Relock Socket & Control — The participants will operate the test socket in one of two test conditions: (1) release/relock mechanisms enabled and (2) release/relock mechanisms disabled. Participants will test each of the two conditions in a random order, out of lab, with no structured protocol. Tests will determine how the novel release/relock mechanisms compare against traditional socket release methods.
  Arms: Release/Relock Socket & Control

SUMMARY:
The goal of the research is to create and evaluate a new technology for management of daily residual limb fluid volume fluctuation.

DETAILED DESCRIPTION:
Limb fluid volume changes that can occur in the residual limb of a lower-limb amputee can result in changes in socket fit that lead to discomfort, skin injuries, and reduced mobility. It is known that limb fluid volume fluctuations can be reduced for some people by intermittently removing (doffing) the socket throughout the day. It is believed that partially doffing the socket may have a similar benefit, and could be made more convenient thereby promoting easier compliance for prosthetic users.

The goal of the research is to create and evaluate a new technology for management of daily residual limb fluid volume fluctuation. The technology enables partial doffing through the release and relock of a socket panel and the prosthetic pin used to hold the limb in place. The expected outcomes are an enhanced understanding of how socket adjustments after activity facilitate limb fluid volume recovery, subsequent fluid retention, and improved socket fit.

ELIGIBILITY:
Inclusion Criteria:

* Had trans-tibial amputation at least 18 months prior to enrollment
* Regularly wear a definitive prosthesis for at least 7 hours per week
* Have a residual limb length of at least 9 cm
* K2 or higher MFCL
* Able to walk continuously with a prosthesis for at least 2 minutes at a time
* Sit, stand, and negotiate a step of 5.0 cm

Participants involved remotely will have to meet the following inclusion criteria:

* Have a spare prosthesis
* No cognitive issues
* Good hand dexterity and strength (not frail)
* Capable of communication over a video Zoom conference call.

Exclusion Criteria:

* Current presence of skin breakdown
* Unable to satisfy inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Limb Volume | Change from baseline period (no release/relock) to test period (release/relock), commonly each 1 hour long and separated by a seated period of approximately 30 minutes
  Limb volume fluctuations will be measured in real-time as socket release/relock strategies are tested. This will be accomplished using a portable bioimpedance device with thin sticky electrodes that are placed on the residual limb. Specifically, the change in limb volume will be assessed from a baseline period where no socket adjustments are made to another period within the same test session where socket adjustments are made.
Prosthesis Evaluation Questionnaire (PEQ) | Administered following out of lab testing, after at least 2 days using the test socket in out-of-lab environments.
  Participants will be asked to fill out a questionnaire related to their experience using the test socket out of lab in various test configurations. Each question on the PEQ can receive a score form 0 to 100, with higher scores indicating greater satisfaction.
PROMIS-Fatigue | Administered following out of lab testing, after at least 2 days using the test socket in out-of-lab environments.
  Participants will be asked to fill out a questionnaire related to their experience using the test socket out of lab in various test configurations. Each PROMIS-Fatigue question asks participants to rank on a scale from 1 to 5 (categorical options), with higher scores indicating greater level of fatigue.
Socket Comfort Score (SCS) | Administered following out of lab testing, after at least 2 days using the test socket in out-of-lab environments.
  Participants will be asked to rank their comfort while using the test socket out of lab in various test configurations. The SCS ranges from 0 to 10 (categorical), with higher scores indicating greater level of comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Joan E Sanders, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Bioengineering, Seattle, Washington, United States